CLINICAL TRIAL: NCT02642211
Title: An Evaluation of Intraocular Pressure Reduction Following Phacoemulsification and Manual Small Incision Cataract Surgery: A Randomized Controlled Trial
Brief Title: IOP Changes Associated With SICS and Phako
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Robin, Alan L., M.D. (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SICS_Phaco_1
Record Dates: First submitted 2015-12-19; First posted 2015-12-30 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2015-12

CONDITIONS: Cataract; Glaucoma
MeSH Terms: conditions — Cataract; Glaucoma | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- phako (Active Comparator): eyes receiving phakoemulsification for cataract surgery
  Interventions: Procedure: cataract surgery
- MSICS (Active Comparator): Eyes undergoing manual small incision cataract surgery
  Interventions: Procedure: cataract surgery

INTERVENTIONS:
Procedure: cataract surgery — Eyes (one eye per patient) randomized to either phacoemulsification and intraocular lens insertion or small incision cataract surgery and intraocular lens insertion

SUMMARY:
Prospective randomized trial in patients requiring cataract surgery in which IOP, angle anatomy and other demographic and clinical data are compared. Subjects randomized to both MSICS and phakoemulsification

DETAILED DESCRIPTION:
Prospective, randomized, double masked, parallel assignment clincal trial. Five hundred eyes of 500 participants between 40 - 70 years with normal IOP, gonioscopically open angles and age related cataract. Eyes underwent phacoemulsification or MSICS following a 1:1 randomization and allocation code. Best corrected vision (BCVA), IOP, comprehensive slit lamp evaluation and anterior segment optical coherence tomography (ASOCT) were performed at baseline and at 1, 3 and 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:Age over 40 requiring cataract surgery -

Exclusion Criteria: inability to follow up, lens not suitable for phacoemulsification, prior intraocular surgery, glaucoma

-

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure lowering | 6 months
  intraocular pressure measured with aplanation tonometry

SECONDARY OUTCOMES:
Angle anatomy | 6 months
  OCT changes in angle anatomy

IPD SHARING:
Plan to Share IPD: Yes
plan to share in paper form and at national meetings